CLINICAL TRIAL: NCT00167622
Title: Efficacy and Safety of Preventive Mechanical Ventilation in Adults With Guillain Barré Syndrome
Brief Title: Early Mechanical Ventilation for Guillain Barré Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Versailles (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Djillali Annane, Professor in medicine, University of Versailles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P050103; PS050103
Record Dates: First submitted 2005-09-10; First posted 2005-09-14 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Guillain Barré Syndrome; Acute Respiratory Failure
Keywords: Guillain Barré; Mechanical ventilation, invasive; Mechanical ventilation, non invasive; Pneumonia
MeSH Terms: conditions — Guillain-Barre Syndrome; Pneumonia | interventions — Respiration, Artificial; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Physiotherapy, oxygen as needed
  Interventions: Procedure: physiotherapy and oxygen if needed
- 2 (Experimental): Mechanical ventilation
  Interventions: Procedure: mechanical ventilation

INTERVENTIONS:
Procedure: mechanical ventilation — Non invasive mechanical ventilation at least 6 hours per day - if difficult swallowing, tracheal intubation and invasive mechanical ventilation
  Arms: 2
Procedure: physiotherapy and oxygen if needed — oxygen will be delivered via facial mask whenever needed and physiotherapy
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether early mechanical ventilation can prevent hospital acquired pneumonia in adults with Guillain Barré Syndrome.

DETAILED DESCRIPTION:
Hospital acquired pneumonia is a common and severe complication of Guillain Barré Syndrome. Several factors have been recognized as predictors of respiratory failure in adults with Guillain Barré Syndrome. They include a time from disease onset and patient admission of less seven days, inability to lift head, impaired swallowing and a forced vital capacity of less than 60% of predictive value. We reasonned that early mechanical ventilation may prevent aspiration which is likely the main cause of pneumonia in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Guillain Barré Syndrome
* Age of 18 years old or more
* Inability to lift head
* Time from onset of motor deficit less than 7 days
* Written informed consent

Exclusion Criteria:

* Glasgow coma score of less than 8
* Unstable hemodynamic status
* Current pneumonia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-04; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Rate of hospital acquired pneumonia from randomization to study day 90 | Day 90

SECONDARY OUTCOMES:
Time on a ventilator | Day 90
Intensive care unit lenght of stay | Day 90
Hospital length of stay | Day 90
Tolerance | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Djillali annane, MD, PhD, Study Chair — Raymond Poincaré Hospital, AP-HP
Locations (1):
- Raymond Poincaré Hospital, Garches, France

REFERENCES:
- [Background] Sharshar T, Chevret S, Bourdain F, Raphael JC; French Cooperative Group on Plasma Exchange in Guillain-Barre Syndrome. Early predictors of mechanical ventilation in Guillain-Barre syndrome. Crit Care Med. 2003 Jan;31(1):278-83. doi: 10.1097/00003246-200301000-00044. PMID 12545029
- [Background] Chevrolet JC, Deleamont P. Repeated vital capacity measurements as predictive parameters for mechanical ventilation need and weaning success in the Guillain-Barre syndrome. Am Rev Respir Dis. 1991 Oct;144(4):814-8. doi: 10.1164/ajrccm/144.4.814. PMID 1928954
- [Derived] Melone MA, Heming N, Meng P, Mompoint D, Aboab J, Clair B, Salomon J, Sharshar T, Orlikowski D, Chevret S, Annane D. Early mechanical ventilation in patients with Guillain-Barre syndrome at high risk of respiratory failure: a randomized trial. Ann Intensive Care. 2020 Sep 30;10(1):128. doi: 10.1186/s13613-020-00742-z. PMID 32997260